CLINICAL TRIAL: NCT02645578
Title: Asia Coma Electrical Stimulation Trial: an Asian Multicenter Randomized Controlled Trial to Assess the Efficacy and Safety of Right Median Nerve Stimulation for Traumatic Coma
Brief Title: Asia Coma Electrical Stimulation (the ACES Trial)
Acronym: ACES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: All India Institute of Medical Sciences (Other); JSC National Center for Neurosurgery, Republic of Kazakhstan (Unknown); College of Medical Sciences Teaching Hospital. Nepal (Other)
Responsible Party: Principal Investigator, Guoyi Gao, Associate professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Renjineuro
Record Dates: First submitted 2015-12-23; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: Coma; traumatic brain injury; median nerve stimulation
MeSH Terms: conditions — Brain Injuries, Traumatic; Coma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RMNS group (Experimental): Focus intervention: right median nerve stimulation plus standard management
  Interventions: Device: Right median nerve stimulation
- Control group (No Intervention): Standard management

INTERVENTIONS:
Device: Right median nerve stimulation — Right median nerve electrical stimulation (RMNS) is administered via a pair of lubricated one-inch square rubber surface electrodes pasted on the volar aspect of the right distal forearm over the median nerve. An electrical neuromuscular stimulator supplied trains of asymmetric biphasic pluses at an amplitude of 20 milliamps with a pulse width of 300 microseconds at 40 Hz for 20 sec/min. The RMNS treatment continues 8 hours per day for two weeks.
  Other Names: RMNS
  Arms: RMNS group

SUMMARY:
This study is a prospective multicenter randomized controlled trial from Asian countries to compare the effect and safety of right median nerve stimulation versus traditional treatment for comatose patients at the early stage following traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a leading cause of mortality and morbidity and one of the greatest unmet needs in public health. The most severe injury can lead to a poor outcome and prolonged coma of the victims. It is estimated that ten to fifteen percent of the severe TBI patients are discharged in a prolonged coma or a vegetative state. However, no treatment measure to data has been proven robustly to alter the pace of recovery or improve neurological outcome of the comatose patients following TBI.

Although right median nerve electrical stimulation (RMNS) has been used clinically for more than two decades, no strong evidence of efficacy was generated because of the limitations in the past trials including a small sample size or the inappropriate study design. In the present study, a multicenter research network with inclusion of neurotrauma centers from China, India, Nepal and Kazakhstan was established with the aim to validate the efficacy and safety of a promising intervention strategy for traumatic coma at early stage. Since RMNS is a simple, inexpensive, noninvasive technique with a good safety profile, our study will probably add more evidence to the treatment of traumatic coma in Asian countries.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed history of closed traumatic brain injury 10 days before enrollment
* A Glasgow coma scale (GCS) score of 4-8 or the motor part less than 5 if the patient received tracheotomy.
* 18-65 years of age

Exclusion Criteria:

* Unstable vital signs
* Have a history of severe cardiac arrhythmias, implanted pacemaker, as well as seizures
* Pregnancy
* No informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients returning consciousness | Within six months after injury
  The term "consciousness" is defined when the patient shows objective ability to respond to verbal commands.

SECONDARY OUTCOMES:
Duration of unconsciousness | Within six months after injury
  This outcome is defined as the time between trauma and objective recovery of the ability to respond to verbal commands
Adverse events | Within six months post injury
  The potential adverse events include but not limited to seizures, intracranial bleeding, increased sympathetic activity and so on.
Glasgow Coma Scale (GCS) | 28 days post injury
Coma Recovery Scale-Revised (CRS-R) | six months post injury
Disability Rating Scale (DRS) | six months post injury
Full Outline of UnResponsiveness scale(FOUR) | 28 days post injury

CONTACTS AND LOCATIONS:
Overall Officials: Jiyao Jiang, Study Chair — RenJi Hospital; Junfeng Feng, Study Director — RenJi Hospital; Guoyi Gao, Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lei J, Wang L, Gao G, Cooper E, Jiang J. Right Median Nerve Electrical Stimulation for Acute Traumatic Coma Patients. J Neurotrauma. 2015 Oct 15;32(20):1584-9. doi: 10.1089/neu.2014.3768. Epub 2015 May 7. PMID 25664378
- [Background] Cooper EB, Scherder EJ, Cooper JB. Electrical treatment of reduced consciousness: experience with coma and Alzheimer's disease. Neuropsychol Rehabil. 2005 Jul-Sep;15(3-4):389-405. doi: 10.1080/09602010443000317. PMID 16350980
- [Background] Liu JT, Wang CH, Chou IC, Sun SS, Koa CH, Cooper E. Regaining consciousness for prolonged comatose patients with right median nerve stimulation. Acta Neurochir Suppl. 2003;87:11-4. doi: 10.1007/978-3-7091-6081-7_3. PMID 14518515
- [Background] Cooper EB, Cooper JB. Electrical treatment of coma via the median nerve. Acta Neurochir Suppl. 2003;87:7-10. doi: 10.1007/978-3-7091-6081-7_2. PMID 14518514
- [Background] Peri CV, Shaffrey ME, Farace E, Cooper E, Alves WM, Cooper JB, Young JS, Jane JA. Pilot study of electrical stimulation on median nerve in comatose severe brain injured patients: 3-month outcome. Brain Inj. 2001 Oct;15(10):903-10. doi: 10.1080/02699050110065709. PMID 11595086
- [Derived] Wu X, Xie L, Lei J, Yao J, Li J, Ruan L, Hong J, Zheng G, Cheng Y, Long L, Wang J, Huang C, Xie Q, Zhang X, He J, Yu X, Lv S, Sun Z, Liu D, Li X, Zhu J, Yang X, Wang D, Bao Y, Maas AIR, Menon D, Xue Y, Jiang J, Feng J, Gao G; ACES Participants. Acute traumatic coma awakening by right median nerve electrical stimulation: a randomised controlled trial. Intensive Care Med. 2023 Jun;49(6):633-644. doi: 10.1007/s00134-023-07072-1. Epub 2023 May 13. PMID 37178149
- [Derived] Wu X, Zhang C, Feng J, Mao Q, Gao G, Jiang J. Right median nerve electrical stimulation for acute traumatic coma (the Asia Coma Electrical Stimulation trial): study protocol for a randomised controlled trial. Trials. 2017 Jul 10;18(1):311. doi: 10.1186/s13063-017-2045-x. PMID 28693604